CLINICAL TRIAL: NCT00274716
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of MK0736 and MK0916 in Hypertensive Patients
Brief Title: Safety and Efficacy of MK0736 & MK0916 in Patients With Hypertension (High Blood Pressure)(0736-003)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0736-003; 2006_004
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Results first posted 2014-02-14 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-06

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — MK-0916

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- High BMI:MK-0736 2mg→Placebo (Experimental): Participants administered MK-0736 2mg tablet once daily for 12 weeks (Phase A) then administered placebo once daily for 12 weeks (Phase B)
  Interventions: Drug: MK0736; Drug: Placebo
- High BMI:MK-0736 7mg→Placebo (Experimental): Participants administered MK-0736 7mg tablet once daily for 12 weeks (Phase A) then administered placebo once daily for 12 weeks (Phase B)
  Interventions: Drug: MK0736; Drug: Placebo
- High BMI:MK-0916 6mg→MK-0916 6mg (Experimental): Participants administered MK-0916 6mg tablet once daily in both Phase A (12 weeks) and Phase B (12 weeks)
  Interventions: Drug: MK0916
- High BMI:Placebo→Placebo (Placebo Comparator): Participants administered placebo tablet once daily in both Phase A (12 weeks) and Phase B (12 weeks)
  Interventions: Drug: Placebo
- Low BMI:MK-0916 6mg→MK-0916 6mg (Experimental): Participants administered MK-0916 6mg tablet once daily in both Phase A (12 weeks) and Phase B (12 weeks)
  Interventions: Drug: MK0916
- Low BMI:Placebo→Placebo (Placebo Comparator): Participants administered placebo tablet once daily in both Phase A (12 weeks) and Phase B (12 weeks)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MK0736
  Arms: High BMI:MK-0736 2mg→Placebo; High BMI:MK-0736 7mg→Placebo
Drug: MK0916
  Arms: High BMI:MK-0916 6mg→MK-0916 6mg; Low BMI:MK-0916 6mg→MK-0916 6mg
Drug: Placebo
  Arms: High BMI:MK-0736 2mg→Placebo; High BMI:MK-0736 7mg→Placebo; High BMI:Placebo→Placebo; Low BMI:Placebo→Placebo

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of two investigational drugs (MK-0736 and MK-0916) in lowering blood pressure and body weight in patients with hypertension (high blood pressure).

This is an early phase trial and some specific protocol information is proprietary and not publicly available at this time. (Full information is available to trial participants).

DETAILED DESCRIPTION:
Participants enrolled in the study will be separated into 2 strata based on baseline body mass index (BMI) assessments prior to being randomly assigned to study treatment. Study will include a 24-week treatment period comprised of 2 phases, A and B, each of which will 12 weeks in duration.

ELIGIBILITY:
Inclusion Criteria:

* Hypertension systolic blood pressure (SBP) </= 160mm Hg and diastolic blood pressure (DBP): 90-105mm Hg

Exclusion Criteria:

* Pre-menopausal women
* patients currently taking more than two (2) blood pressure lowering medications
* Body Mas Index (BMI)>40 kg/m2 (morbidly obese patients)
* History of Alcohol abuse (<3 Years)
* History of diabetes,chronic kidney disease, Active liver disease, recent heart attack or stroke

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2005-11; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Shah S, Hermanowski-Vosatka A, Gibson K, Ruck RA, Jia G, Zhang J, Hwang PM, Ryan NW, Langdon RB, Feig PU. Efficacy and safety of the selective 11beta-HSD-1 inhibitors MK-0736 and MK-0916 in overweight and obese patients with hypertension. J Am Soc Hypertens. 2011 May-Jun;5(3):166-76. doi: 10.1016/j.jash.2011.01.009. Epub 2011 Mar 21. PMID 21419745

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrolled participants were divided into 2 strata: higher body mass index (BMI) (27 kg/m^2≤BMI<41 kg/m^2) and lower BMI (20 kg/m^2≤BMI<27 kg/m^2) prior to being randomly assigned study treatment. Data from High BMI groups were to be utilized in the primary and secondary analyses; data from low BMI groups were to be utilized in exploratory analyses.
Period: Phase A
Arm/Group | High BMI:MK-0736 2mg→Placebo | High BMI:MK-0736 7mg→Placebo | High BMI:MK-0916 6mg→MK-0916 6mg | High BMI:Placebo→Placebo | Low BMI:MK-0916 6mg→MK-0916 6mg | Low BMI:Placebo→Placebo
Started | 54 | 54 | 52 | 51 | 19 | 19
Completed | 43 | 44 | 44 | 42 | 16 | 15
Not Completed | 11 | 10 | 8 | 9 | 3 | 4
Not completed — Other non-reported reason | 4 | 2 | 1 | 2 | 0 | 1
Not completed — Participant moved | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Site Terminated | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Met criteria for discontinuation | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 1 | 3 | 0 | 1
Not completed — Adverse Event | 2 | 3 | 3 | 0 | 2 | 0
Not completed — Completed but did not enter Phase B | 1 | 2 | 2 | 2 | 1 | 1
Period: Phase B
Arm/Group | High BMI:MK-0736 2mg→Placebo | High BMI:MK-0736 7mg→Placebo | High BMI:MK-0916 6mg→MK-0916 6mg | High BMI:Placebo→Placebo | Low BMI:MK-0916 6mg→MK-0916 6mg | Low BMI:Placebo→Placebo
Started | 43 | 44 | 44 | 42 | 16 | 15
Completed | 42 | 40 | 41 | 41 | 16 | 14
Not Completed | 1 | 4 | 3 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 2 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Participant moved | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Other non-reported reason | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- High BMI:MK-0916 6mg→MK-0916 6mg: Participants who received MK-0916 6 mg in Phase A and continued on MK-0916 6 mg for 12 weeks in Phase B
- Total: Total of all reporting groups
Arm/Group | High BMI:MK-0736 2mg→Placebo | High BMI:MK-0736 7mg→Placebo | High BMI:MK-0916 6mg→MK-0916 6mg | High BMI:Placebo→Placebo | Low BMI:MK-0916 6mg→MK-0916 6mg | Low BMI:Placebo→Placebo | Total
Number analyzed (Participants) | 54 | 54 | 52 | 51 | 19 | 19 | 249
Age, Customized [Number; unit: Participants]
  21 to 30 years | 0 | 1 | 0 | 1 | 0 | 0 | 2
  31 to 40 years | 3 | 3 | 0 | 6 | 0 | 0 | 12
  41 to 50 years | 10 | 17 | 20 | 14 | 6 | 4 | 71
  51 to 60 years | 26 | 20 | 20 | 17 | 9 | 9 | 101
  61 to 70 years | 14 | 12 | 12 | 13 | 4 | 6 | 61
  >70 years | 1 | 1 | 0 | 0 | 0 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 17 | 20 | 13 | 6 | 10 | 96
  Male | 24 | 37 | 32 | 38 | 13 | 9 | 153

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough Sitting Diastolic Blood Pressure (SiDBP) at Week 12 in Participants With Higher Body Mass Indices (BMI)
Description: Sitting diastolic blood pressure measured in triplicate at baseline and after 12 weeks of study drug administration. Mean value of the 3 measurements at the 2 timepoints was recorded.
Time Frame: Baseline and Week 12 (end of Phase A)
Population: Higher BMI participants in the All Patients Treated (APT) Population, which included all randomized participants who had valid efficacy measurements at baseline and at least once during the double-blind treatment period. The MK-0916 6.0 mg and Placebo Low BMI groups were not included in the planned analysis for this endpoint.
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- MK-0736 2.0 mg High BMI: Participants administered MK-0736 2.0 mg tablet once daily for 12 weeks
- MK-0736 7.0 mg High BMI: Participants administered MK-0736 7.0 mg tablet once daily for 12 weeks
- MK-0916 6.0 mg High BMI: Participants administered MK-0916 6.0 mg tablet once daily for 12 weeks
- Placebo High BMI: Participants administered placebo tablet once daily for 12 weeks
Arm/Group | MK-0736 2.0 mg High BMI | MK-0736 7.0 mg High BMI | MK-0916 6.0 mg High BMI | Placebo High BMI
Number analyzed (Participants) | 53 | 52 | 49 | 51
mm Hg | -4.2 (7.3) | -2.4 (8.1) | -3.1 (7.9) | -0.2 (8.7)
Statistical Analysis 1: Comparison: MK-0736 7.0 mg High BMI vs Placebo High BMI; Test type: Superiority or Other; p = 0.157, ANCOVA; Treatment group and ambulatory blood pressure measurement (ABPM; yes or no) as class variables and baseline mean trough SiDBP as a continuous variable; Mean Difference (Final Values) = -2.2, 95% CI 2-sided [-5.3 to 0.9], Standard Error of Mean 1.6
Statistical Analysis 2: Comparison: MK-0736 2.0 mg High BMI vs Placebo High BMI; Test type: Superiority or Other; p = 0.010, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.1, 95% CI 2-sided [-7.1 to -1.0], Standard Error of Mean 1.5
Statistical Analysis 3: Comparison: MK-0916 6.0 mg High BMI vs Placebo High BMI; Test type: Superiority or Other; p = 0.042, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.2, 95% CI 2-sided [-6.4 to -0.1], Standard Error of Mean 1.6
Statistical Analysis 4: Comparison: MK-0736 7.0 mg High BMI vs MK-0916 6.0 mg High BMI; Test type: Superiority or Other; p = 0.517, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.0, 95% CI 2-sided [-2.1 to 4.1], Standard Error of Mean 1.6
Statistical Analysis 5: Comparison: MK-0736 2.0 mg High BMI vs MK-0916 6.0 mg High BMI; Test type: Superiority or Other; p = 0.602, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-3.9 to 2.3], Standard Error of Mean 1.6

2. Secondary Outcome: Change From Baseline in Trough Sitting Systolic Blood Pressure (SiSBP) at Week 12 in Participants With Higher Body Mass Indices (BMI)
Description: Sitting systolic blood pressure measured in triplicate at baseline and after 12 weeks of study drug administration. Mean trough value of the 3 measurements at the 2 timepoints was recorded.
Time Frame: Baseline and Week 12 (end of Phase A)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | MK-0736 2.0 mg High BMI | MK-0736 7.0 mg High BMI | MK-0916 6.0 mg High BMI | Placebo High BMI
Number analyzed (Participants) | 53 | 52 | 49 | 51
mm Hg | -3.5 (13.2) | -4.2 (12.9) | -3.2 (11.3) | 0.7 (12.2)
Statistical Analysis 1: Comparison: MK-0736 7.0 mg High BMI vs Placebo High BMI; Test type: Superiority or Other; p = 0.046, ANCOVA; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = -4.9, 95% CI 2-sided [-9.7 to -0.1], Standard Error of Mean 2.4
Statistical Analysis 2: Comparison: MK-0736 2.0 mg High BMI vs Placebo High BMI; Test type: Superiority or Other; p = 0.108, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.9, 95% CI 2-sided [-8.7 to 0.9], Standard Error of Mean 2.4
Statistical Analysis 3: Comparison: MK-0916 6.0 mg High BMI vs Placebo High BMI; Test type: Superiority or Other; p = 0.099, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.1, 95% CI 2-sided [-9.0 to 0.8], Standard Error of Mean 2.5
Statistical Analysis 4: Comparison: MK-0736 7.0 mg High BMI vs MK-0916 6.0 mg High BMI; Test type: Superiority or Other; p = 0.752, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-5.7 to 4.1], Standard Error of Mean 2.5
Statistical Analysis 5: Comparison: MK-0736 2.0 mg High BMI vs MK-0916 6.0 mg High BMI; Test type: Superiority or Other; p = 0.941, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-4.7 to 5.0], Standard Error of Mean 2.5

3. Secondary Outcome: Change From Baseline in Body Weight (kg) at Week 12 in Participants With Higher BMI
Description: Weight was measured in duplicate (2 measurements) at baseline and after 12 weeks of study drug administration. The mean of the 2 values at each assessment was used in analysis.
Time Frame: Baseline and Week 12 (end of Phase A)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | MK-0736 2.0 mg High BMI | MK-0736 7.0 mg High BMI | MK-0916 6.0 mg High BMI | Placebo High BMI
Number analyzed (Participants) | 54 | 52 | 50 | 50
kg | -0.6 (1.8) | -0.9 (2.0) | -1.2 (1.8) | 0.5 (1.9)
Statistical Analysis 1: Comparison: MK-0736 7.0 mg High BMI vs Placebo High BMI; Test type: Superiority or Other; p < 0.001, ANCOVA; Treatment group and ambulatory blood pressure measurement (ABPM; yes or no) as class variables and baseline weight as a continuous variable; Median Difference (Final Values) = -1.4, 95% CI 2-sided [-2.2 to -0.7], Standard Error of Mean 0.4
Statistical Analysis 2: Comparison: MK-0736 2.0 mg High BMI vs Placebo High BMI; Test type: Superiority or Other; p = 0.003, ANCOVA; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-1.9 to -0.4], Standard Error of Mean 0.4
Statistical Analysis 3: Comparison: MK-0916 6.0 mg High BMI vs Placebo High BMI; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-2.4 to -1.0], Standard Error of Mean 0.4
Statistical Analysis 4: Comparison: MK-0736 7.0 mg High BMI vs MK-0916 6.0 mg High BMI; Test type: Superiority or Other; p = 0.462, ANCOVA; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-0.5 to 1.0], Standard Error of Mean 0.4
Statistical Analysis 5: Comparison: MK-0736 2.0 mg High BMI vs MK-0916 6.0 mg High BMI; Test type: Superiority or Other; p = 0.118, ANCOVA; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-0.2 to 1.3], Standard Error of Mean 0.4

4. Secondary Outcome: Change From Baseline in Waist Circumference at Week 12 in Participants With Higher BMI
Description: Waist circumference measured in cm at baseline and after 12 weeks of study drug administration
Time Frame: Baseline and Week 12 (end of Phase A)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | MK-0736 2.0 mg High BMI | MK-0736 7.0 mg High BMI | MK-0916 6.0 mg High BMI | Placebo High BMI
Number analyzed (Participants) | 47 | 50 | 49 | 44
cm | -1.9 (4.9) | -0.9 (2.9) | -0.3 (4.9) | 1.2 (6.1)
Statistical Analysis 1: Comparison: MK-0736 7.0 mg High BMI vs Placebo High BMI; Test type: Superiority or Other; p = 0.059, ANCOVA; Treatment group and ambulatory blood pressure measurement (ABPM; yes or no) as class variables and baseline waist as a continuous variable; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-3.7 to 0.1], Standard Error of Mean 0.9
Statistical Analysis 2: Comparison: MK-0736 2.0 mg High BMI vs Placebo High BMI; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -3.6, 95% CI 2-sided [-5.5 to -1.7], Standard Error of Mean 1.0
Statistical Analysis 3: Comparison: MK-0916 6.0 mg High BMI vs Placebo High BMI; Test type: Superiority or Other; p = 0.136, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-3.3 to 0.5], Standard Error of Mean 0.9
Statistical Analysis 4: Comparison: MK-0736 7.0 mg High BMI vs MK-0916 6.0 mg High BMI; Test type: Superiority or Other; p = 0.686, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-2.2 to 1.4], Standard Error of Mean 0.9
Statistical Analysis 5: Comparison: MK-0736 2.0 mg High BMI vs MK-0916 6.0 mg High BMI; Test type: Superiority or Other; p = 0.022, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -2.2, 95% CI 2-sided [-4.0 to -0.3], Standard Error of Mean 0.9

5. Secondary Outcome: Percent Change From Baseline in Low Density Lipoprotein Cholesterol (LDL-C) at Week 12 in Participants With Higher Body Mass Indices (BMI)
Description: LDL-C was calculated by the method of Friedewald equation at baseline and after 12 weeks of study drug administration.
Time Frame: Baseline and Week 12 (end of Phase A)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | MK-0736 2.0 mg High BMI | MK-0736 7.0 mg High BMI | MK-0916 6.0 mg High BMI | Placebo High BMI
Number analyzed (Participants) | 49 | 50 | 44 | 45
percentage change | -1.0 (23.3) | -5.2 (20.4) | 4.5 (23.0) | 5.7 (30.8)
Statistical Analysis 1: Comparison: MK-0736 7.0 mg High BMI vs Placebo High BMI; Test type: Superiority or Other; p = 0.005, ANCOVA; Treatment group and ambulatory blood pressure measurement (ABPM; yes or no) as class variables and baseline LDL-C as a continuous variable; Mean Difference (Final Values) = -12.3, 95% CI 2-sided [-20.8 to -3.7], Standard Error of Mean 4.3
Statistical Analysis 2: Comparison: MK-0736 2.0 mg High BMI vs Placebo High BMI; Test type: Superiority or Other; p = 0.066, ANCOVA; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -8.1, 95% CI 2-sided [-16.7 to 0.5], Standard Error of Mean 4.4
Statistical Analysis 3: Comparison: MK-0916 6.0 mg High BMI vs Placebo High BMI; Test type: Superiority or Other; p = 0.319, ANCOVA; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -4.5, 95% CI 2-sided [-13.4 to 4.4], Standard Error of Mean 4.5
Statistical Analysis 4: Comparison: MK-0736 7.0 mg High BMI vs MK-0916 6.0 mg High BMI; Test type: Superiority or Other; p = 0.077, ANCOVA; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -7.8, 95% CI 2-sided [-16.4 to 0.8], Standard Error of Mean 4.4
Statistical Analysis 5: Comparison: MK-0736 2.0 mg High BMI vs MK-0916 6.0 mg High BMI; Test type: Superiority or Other; p = 0.418, ANCOVA; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -3.6, 95% CI 2-sided [-12.2 to 5.1], Standard Error of Mean 4.4

6. Secondary Outcome: Change From Baseline for High Density Lipoprotein Cholesterol (HDL-C) at Week 12 in Participants With Higher BMI
Description: HDL-C measured at baseline and after 12 weeks of study drug administration.
Time Frame: Baseline and Week 12 (end of Phase A)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | MK-0736 2.0 mg High BMI | MK-0736 7.0 mg High BMI | MK-0916 6.0 mg High BMI | Placebo High BMI
Number analyzed (Participants) | 49 | 51 | 47 | 45
Percent change | -1.3 (5.7) | -1.8 (6.7) | 1.6 (6.7) | 1.5 (5.0)
Statistical Analysis 1: Comparison: MK-0736 7.0 mg High BMI vs Placebo High BMI; Test type: Superiority or Other; p = 0.015, ANCOVA; Treatment group and ambulatory blood pressure measurement (ABPM; yes or no) as class variables and baseline HDL-C as a continuous variable; Mean Difference (Final Values) = -6.3, 95% CI 2-sided [-11.3 to -1.2], Standard Error of Mean 2.5
Statistical Analysis 2: Comparison: MK-0736 2.0 mg High BMI vs Placebo High BMI; Test type: Superiority or Other; p = 0.124, ANCOVA; [statistical method as in outcome 6, analysis 1]; Mean Difference (Final Values) = -4.0, 95% CI 2-sided [-9.2 to 1.1], Standard Error of Mean 2.6
Statistical Analysis 3: Comparison: MK-0916 6.0 mg High BMI vs Placebo High BMI; Test type: Superiority or Other; p = 0.429, ANCOVA; [statistical method as in outcome 6, analysis 1]; Mean Difference (Final Values) = 2.1, 95% CI 2-sided [-3.1 to 7.2], Standard Error of Mean 2.6
Statistical Analysis 4: Comparison: MK-0736 7.0 mg High BMI vs MK-0916 6.0 mg High BMI; Test type: Superiority or Other; p = 0.001, ANCOVA; [statistical method as in outcome 6, analysis 1]; Mean Difference (Final Values) = -8.3, 95% CI 2-sided [-13.3 to -3.4], Standard Error of Mean 2.5
Statistical Analysis 5: Comparison: MK-0736 2.0 mg High BMI vs MK-0916 6.0 mg High BMI; Test type: Superiority or Other; p = 0.018, ANCOVA; [statistical method as in outcome 6, analysis 1]; Mean Difference (Final Values) = -6.1, 95% CI 2-sided [-11.1 to -1.1], Standard Error of Mean 2.5

7. Secondary Outcome: Percent Change From Baseline in Triglycerides (TG) at Week 12 in Participants With Higher Body Mass Indices (BMI)
Description: TG measured at baseline and after 12 weeks of study drug administration
Time Frame: Baseline and Week 12 (end of Phase A)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | MK-0736 2.0 mg High BMI | MK-0736 7.0 mg High BMI | MK-0916 6.0 mg High BMI | Placebo High BMI
Number analyzed (Participants) | 49 | 51 | 47 | 45
Percent change | 11.5 (40.3) | 20.1 (54.9) | 11.6 (41.2) | 11.1 (40.2)
Statistical Analysis 1: Comparison: MK-0736 7.0 mg High BMI vs Placebo High BMI; Test type: Superiority or Other; p = 0.587, ANCOVA; Treatment group and ambulatory blood pressure measurement (ABPM; yes or no) as class variables and baseline TG as a continuous variable; Mean Difference (Final Values) = 4.9, 95% CI 2-sided [-12.9 to 22.8], Standard Error of Mean 9.0
Statistical Analysis 2: Comparison: MK-0736 2.0 mg High BMI vs Placebo High BMI; Test type: Superiority or Other; p = 0.562, ANCOVA; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = -5.3, 95% CI 2-sided [-23.5 to 12.8], Standard Error of Mean 9.2
Statistical Analysis 3: Comparison: MK-0916 6.0 mg High BMI vs Placebo High BMI; Test type: Superiority or Other; p = 0.802, ANCOVA; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = 2.3, 95% CI 2-sided [-15.8 to 20.4], Standard Error of Mean 9.2
Statistical Analysis 4: Comparison: MK-0736 7.0 mg High BMI vs MK-0916 6.0 mg High BMI; Test type: Superiority or Other; p = 0.772, ANCOVA; [statistical method as in outcome 7, analysis 1]; Median Difference (Final Values) = 2.6, 95% CI 2-sided [-15.2 to 20.5], Standard Error of Mean 9.0
Statistical Analysis 5: Comparison: MK-0736 2.0 mg High BMI vs MK-0916 6.0 mg High BMI; Test type: Superiority or Other; p = 0.409, ANCOVA; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = -7.6, 95% CI 2-sided [-25.9 to 10.6], Standard Error of Mean 9.2

8. Primary Outcome: Number of Participants Who Reported a Clinical Adverse Event
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR'S product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the SPONSOR'S product, is also an AE. A clinical AE was an AE reported as a result of a clinical examination.
Time Frame: 24 weeks
Population: All Patients as Treated (ApaT) population, defined as all randomized participants who received at least 1 dose of double-blind study therapy.
Measure: Number; unit: Participants
Arm/Group | High BMI:MK-0736 2mg→Placebo | High BMI:MK-0736 7mg→Placebo | High BMI:MK-0916 6mg→MK-0916 6mg | High BMI:Placebo→Placebo | Low BMI:MK-0916 6mg→MK-0916 6mg | Low BMI:Placebo→Placebo
Number analyzed (Participants) | 54 | 54 | 52 | 51 | 19 | 19
Participants | 44 | 39 | 38 | 36 | 16 | 11

9. Primary Outcome: Number of Participants Who Reported a Laboratory Adverse Event
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR'S product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the SPONSOR'S product, is also an AE. A laboratory AE was an AE reported as a result of a laboratory assessment or test.
Time Frame: 24 weeks
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | High BMI:MK-0736 2mg→Placebo | High BMI:MK-0736 7mg→Placebo | High BMI:MK-0916 6mg→MK-0916 6mg | High BMI:Placebo→Placebo | Low BMI:MK-0916 6mg→MK-0916 6mg | Low BMI:Placebo→Placebo
Number analyzed (Participants) | 54 | 54 | 52 | 51 | 19 | 19
Participants | 1 | 2 | 0 | 2 | 0 | 0

10. Primary Outcome: Number of Participants Who Were Discontinued From Study Due to Clinical Adverse Event
Description: as for outcome 8
Time Frame: 24 weeks
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | High BMI:MK-0736 2mg→Placebo | High BMI:MK-0736 7mg→Placebo | High BMI:MK-0916 6mg→MK-0916 6mg | High BMI:Placebo→Placebo | Low BMI:MK-0916 6mg→MK-0916 6mg | Low BMI:Placebo→Placebo
Number analyzed (Participants) | 54 | 54 | 52 | 51 | 19 | 19
Participants | 2 | 3 | 6 | 0 | 2 | 1

11. Primary Outcome: Number of Participants Who Were Discontinued From Study Due to Laboratory Adverse Event
Description: as for outcome 9
Time Frame: 24 weeks
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | High BMI:MK-0736 2mg→Placebo | High BMI:MK-0736 7mg→Placebo | High BMI:MK-0916 6mg→MK-0916 6mg | High BMI:Placebo→Placebo | Low BMI:MK-0916 6mg→MK-0916 6mg | Low BMI:Placebo→Placebo
Number analyzed (Participants) | 54 | 54 | 52 | 51 | 19 | 19
Participants | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | High BMI:MK-0736 2mg→Placebo | High BMI:MK-0736 7mg→Placebo | High BMI:MK-0916 6mg→MK-0916 6mg | High BMI:Placebo→Placebo | Low BMI:MK-0916 6mg→MK-0916 6mg | Low BMI:Placebo→Placebo
Serious Adverse Events (participants affected / at risk) | 2/54 | 1/54 | 2/52 | 1/51 | 2/19 | 1/19
Other Adverse Events (participants affected / at risk) | 40/54 | 39/54 | 37/52 | 37/51 | 16/19 | 11/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High BMI:MK-0736 2mg→Placebo (N=54) | High BMI:MK-0736 7mg→Placebo (N=54) | High BMI:MK-0916 6mg→MK-0916 6mg (N=52) | High BMI:Placebo→Placebo (N=51) | Low BMI:MK-0916 6mg→MK-0916 6mg (N=19) | Low BMI:Placebo→Placebo (N=19)
Abdominal Hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Anaphylactic Reaction (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Meningitis Bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Lichen Sclerosus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | High BMI:MK-0736 2mg→Placebo (N=54) | High BMI:MK-0736 7mg→Placebo (N=54) | High BMI:MK-0916 6mg→MK-0916 6mg (N=52) | High BMI:Placebo→Placebo (N=51) | Low BMI:MK-0916 6mg→MK-0916 6mg (N=19) | Low BMI:Placebo→Placebo (N=19)
Constipation (Gastrointestinal disorders) | 3 | 0 | 3 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 4 | 1 | 0 | 1
Chest Pain (General disorders) | 1 | 3 | 0 | 1 | 1 | 0
Fatigue (General disorders) | 2 | 2 | 3 | 1 | 0 | 1
Oedema Peripheral (General disorders) | 2 | 3 | 2 | 2 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1 | 3 | 1 | 1 | 0
Influenza (Infections and infestations) | 4 | 1 | 1 | 2 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 6 | 3 | 4 | 1 | 1
Sinusitis (Infections and infestations) | 2 | 3 | 3 | 3 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 7 | 11 | 7 | 8 | 2 | 3
Urinary Tract Infection (Infections and infestations) | 3 | 0 | 2 | 2 | 0 | 2
Viral Infection (Infections and infestations) | 1 | 0 | 4 | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 6 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 3 | 5 | 3 | 0 | 0
Headache (Nervous system disorders) | 10 | 10 | 15 | 12 | 3 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 1 | 0 | 1 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0
Blepharospasm (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 1 | 0 | 0 | 0 | 1 | 0
Change Of Bowel Habit (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 1 | 2 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 2 | 1 | 1 | 0
Lip Swelling (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 1
Influenza Like Illness (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Oral Herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 1 | 0 | 4 | 0
Tooth Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0
Fluid Retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 2 | 0 | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 2 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 1 | 2 | 2 | 1 | 0 | 1
Sinus Headache (Nervous system disorders) | 0 | 2 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Postmenopausal Haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 1 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hot Flush (Vascular disorders) | 0 | 1 | 1 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication guidelines.